CLINICAL TRIAL: NCT04340323
Title: A Randomized Interventional Parallel Study to Evaluate the Effect of Pelvic Floor Muscle Training With Stabilization Exercises of High and Low Intensity in Women With Stress Urinary Incontinence - the PELSTAB Study
Brief Title: The Effect of Pelvic Floor Muscle Training With Stabilization Exercises With Various Intensity in Women With Stress Urinary Incontinence
Acronym: PELSTAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pavol Jozef Safarik University (Other)
Responsible Party: Principal Investigator, Peter Urdzik, Faculty of Medicine, Pavol Jozef Safarik University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3545/2020/ODDZ-06621
Record Dates: First submitted 2020-04-03; First posted 2020-04-09 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary incontinence;; 2D/3D ultrasound; Pelvic floor muscle training
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A-intensive exercise group (Experimental): Dosage of intensive exercise group - 12 weeks, five times a week for 30 minutes per day; five times with education by a physiotherapist, followed by continuation at home.
  PFMT with lumbopelvic stabilization. Exercise up to five times a week for up to 30 minutes per day, after initial training with a physiotherapist.
  1. Educating probands about anatomy, physiology and pelvic floor muscle function.
  2. Training of pelvic floor muscles in different positions.
  3. Training of pelvic floor muscles with six stabilization exercises - activation of deep trunk muscles.
  Interventions: Other: Pelvic Floor Muscle Training (PFMT)
- Group B-low-intensity exercise group (Active Comparator): Dosage of low-intensity exercise group - 12 weeks, twice a week for 15 minutes per day; five times with physiotherapist education, followed by continuation at home.
  PFMT with lumbopelvic stabilization. Exercise up to five times a week for up to 30 minutes per day, after initial training with a physiotherapist.
  1. Educating probands about anatomy, physiology and pelvic floor muscle function.
  2. Training of pelvic floor muscles in different positions.
  3. Training of pelvic floor muscles with six stabilization exercises - activation of deep trunk muscles.
  Interventions: Other: Pelvic Floor Muscle Training (PFMT)

INTERVENTIONS:
Other: Pelvic Floor Muscle Training (PFMT) — The method of first choice in SUI treatment according to the International Continence Society (ICS) is training of the pelvic floor muscles. Pelvic floor muscle training (PFMT) is a method based on scientific evidence, defined by the ICS as repeated selective voluntary contraction and relaxation of specific pelvic floor muscles. It is important to train the strength and endurance of the pelvic floor muscles but also their relaxation (Abrams, 2018; Arnold, 2014; Bo, 2013).

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of high- and low-intensity PFMT with stabilization exercises in women with SUI

DETAILED DESCRIPTION:
This is a randomized interventional parallel study to evaluate the effect of PFMT with stabilization exercises of high and low intensity in women with SUI

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent
2. Over 18 years old and experiencing uncomplicated SUI
3. Score on the International Consultation on Urinary Incontinence Questionnaire of ≥ 6 points
4. Symptoms of urinary incontinence for at least three consecutive months
5. Degree of pelvic organ prolapse, stage ≤ 2
6. Willingness to accept the randomization process and fully participate in tests

Exclusion Criteria:

1. History of anti-incontinence surgery in the past 12 months
2. History of pelvic prolapse repair or urethral surgery in the past 12 months
3. History of PFMT in the past 12 months
4. History of interstitial cystitis or bladder-related pain
5. Chronic severe constipation
6. Clinically significant renal or hepatic impairment
7. Clinically significant heart impairment
8. Pregnant, lactating or actively trying to become pregnant
9. Positive urinary tract infection
10. Use of rehabilitation aids (pessaries, urethral plugs, vaginal beads, etc.)
11. Insufficient understanding of pelvic floor exercises and/or omitting exercises
12. Incomplete questionnaire
13. Refusal to participate in the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Change in incontinence episode frequency (IEF) over one week. | change in incontinence episode frequency over 12 weeks of treatment
  Change in the number of urinary leakages during the day, measured by the voiding diary.

SECONDARY OUTCOMES:
Change in performance and endurance of pelvic floor muscles | Change in performance and endurance of pelvic floor muscles over 12 weeks of treatment
  Performance on five-degree scale of 0-5 is used (no contraction, weak contraction, normal contraction, strong contraction, very strong contraction).
  Endurance - the patient is requested to perform a maximum voluntary contraction of the pelvic floor and the contraction weakening time is measured. Time is given in seconds, for a maximum of 10 seconds.
Change in hiatal area (HA, in cm2) during the Valsalva manoeuvre, assessed by 3D ultrasound | Change in hiatal area (HA, in cm2) during the Valsalva manoeuvre, assessed by 3D ultrasound over 12 weeks of treatment
  Examination will be carried out using a ultrasound console, volume contrast imaging software and a 3D/4D 4-8 MHz probe in the midsagittal plane. Examination will take place with an empty bladder in the lithotomy position. The probe will be placed longitudinally on the perineum. A 3D image will be taken at rest, at maximum contraction and at the Valsalva manoeuvre. The amount of hiatial space at the Valsalva manoeuvre will be measured in cm2.
Change in incontinence quality of life | Change in incontinence quality of life over 12 weeks of treatment
  Urinary Incontinence Quality of Life Scale (I-QoL)
  The I-QoL is composed of three subscales (avoidance and limiting behaviour; psychosocial impact; social embarrassment) and comprises 22 questions with a total score in the range from 0 (worst quality of life) to 100 (best quality of life).
Change in patient global impression | Change in patient global impression over 12 weeks of treatment
  Patient Global Impression of Improvement Scale (PGI-I)
  The PGI-I evaluates the status of urination problems compared to the patient's condition before treatment in the study. Patient impressions are evaluated according to the following scores: 1, much better; 2, quite better; 3, a little better; 4, no change; 5, a little worse; 6, a lot worse; 7, definitely worse.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Urdzik, prof.MD,PhD, Principal Investigator — Pavol Jozef Safarik University, Faculty of Medicine
Locations (1):
- Pavol Jozef Safarik University, Faculty of Medicine, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322
- [Derived] Hagovska M, Urdzik P, Svihra J. A randomized interventional parallel study to evaluate the effect of pelvic floor muscle training with stabilization exercises of high and low intensity in women with stress urinary incontinence: The PELSTAB study. Medicine (Baltimore). 2020 Jul 17;99(29):e21264. doi: 10.1097/MD.0000000000021264. PMID 32702912